CLINICAL TRIAL: NCT00484341
Title: NGR016: Randomized Phase II Study Evaluating Two Doses of NGR-hTNF Administered Either as Single Agent or in Combination With Doxorubicin in Patients With Advanced Soft Tissue Sarcoma (STS)
Brief Title: Phase II Study of NGR-hTNF in Combination With Doxorubicin in Patients Affected by Soft Tissue Sarcomas.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGR016; 2010-018851-88 (EudraCT Number)
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Adult Soft Tissue Sarcoma
Keywords: NGR-hTNF; Doxorubicin; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: low-dose NGR-hTNF (Experimental): 0.8 mcg/m² of NGR-hTNF
  Interventions: Drug: low-dose NGR-hTNF
- B: high-dose NGR-hTNF (Experimental): 45 mcg/m² of NGR-hTNF
  Interventions: Drug: high-dose NGR-hTNF
- C: low-dose NGR-hTNF + doxorubicin (Experimental): 0.8 mcg/m² of NGR-hTNF + doxorubicin
  Interventions: Drug: low-dose NGR-hTNF; Drug: Doxorubicin
- D: high-dose NGR-hTNF + doxorubicin (Experimental): 45 mcg/m² of NGR-hTNF + doxorubicin
  Interventions: Drug: high-dose NGR-hTNF; Drug: Doxorubicin

INTERVENTIONS:
Drug: low-dose NGR-hTNF — NGR-hTNF: 0.8 mcg/m² as 60-minutes intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs
  Other Names: NGR-hTNF
  Arms: A: low-dose NGR-hTNF; C: low-dose NGR-hTNF + doxorubicin
Drug: high-dose NGR-hTNF — NGR-hTNF: 45 mcg/m² as 60-minutes intravenous infusion every week until confirmed evidence of disease progression or unacceptable toxicity occurs
  Other Names: NGR-hTNF
  Arms: B: high-dose NGR-hTNF; D: high-dose NGR-hTNF + doxorubicin
Drug: Doxorubicin — Doxorubicin: 60 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion) on day 1 every 3 weeks for a maximum of 6 cycles or until cumulative dose of 550 mg/m²
  Arms: C: low-dose NGR-hTNF + doxorubicin; D: high-dose NGR-hTNF + doxorubicin

SUMMARY:
The main objective of the trial is to document the preliminary antitumor activity of two doses of NGR-hTNF administered either alone or in combination with doxorubicin in locally advanced or metastatic soft-tissue sarcoma (STS) patients untreated or previously treated with one or more prior systemic regimen.

DETAILED DESCRIPTION:
Considering the safety/toxicity profile of NGR-hTNF characterized by mild-to-moderate constitutional symptoms when given either every three weeks or weekly both at low (0.8 µg/m^2) and high dose (45 µg/m^2); the reversibility of these adverse events generally occurring only during the infusion time; the absence of overlapping toxicities with chemotherapeutic agents; and the safety and preliminary antitumor activity observed in phase Ib trial with doxorubicin, seems justified to evaluate in a randomized 4-arm phase II trial the preliminary antitumor activity of two doses of NGR-hTNF (0.8 µg/m^2 and 45 µg/m^2) administered weekly either alone or in combination with a standard dose of doxorubicin (60 mg/m^2 every three weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Histologically-proven, locally advanced, or metastatic STS (excluding extraosseus Ewing sarcoma)
* Patients not amenable to surgery, radiotherapy, or combined-modality therapy with curative intent
* Patients untreated or previously treated with one or more systemic regimen
* ECOG Performance status 0-2 (Appendix A)
* At least one untreated (not previously irradiated) target lesion that could be measured in one dimension, according to RECIST criteria
* A life expectancy of 12 weeks or more
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils > 1.5 x 109/L and platelets > 100 x 109/L
  * Bilirubin < 1.5 x ULN
  * AST and/or ALT < 2.5 x ULN in absence of liver metastasis or < 5 x ULN in presence of liver metastasis
  * Serum creatinine < 1.5 x ULN
  * Creatinine clearance (estimated according to Cockcroft-Gault formula) ≥ 50 ml/min
* Patients may have had prior treatment providing the following conditions are met before treatment start:

  * Surgery and radiation therapy: wash-out period of 14 days
  * Systemic therapy: wash-out period of 21 days
  * Patients must give written informed consent

Exclusion Criteria:

* Patients may not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six (6) months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* LVEF < 55% (only for patients candidate for doxorubicin treatment)
* Uncontrolled hypertension
* Prolonged QTc interval (congenital or acquired) > 450 ms
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., primary brain tumor, any brain metastasis, seizure not controlled with standard medical therapy) or history of stroke
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction or contraindications to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of child-bearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | every 6-12 weeks
  Defined as the time from the date of randomization until disease progression, or death

SECONDARY OUTCOMES:
Safety and Toxicity according to NCI-CTCAE criteria (version 4.02) | during the study
  To evaluate safety and toxicity profile related to NGR-hTNF
Duration of Disease Control | every 6-12 weeks
  Measured from the date of randomization until disease progression, or death due to any cause
Overall survival (OS) | every 6-12 weeks
  Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive
Response rate | every 6-12 weeks
  Measured both according to RECIST criteria and by FDG-PET
Tumor response | every 6-12 weeks
  Evaluated by a centralized review of changes in tumor density on CT scan and/or perfusion MRI

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (7):
- France (2):
  - Centre Leon Berard, Lyon
  - Institut de Cancérologie Gustave Roussy, Villejuif
- Italy (4):
  - Istituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan
  - IRCCS Policlinico S. Matteo, Pavia
  - Università Campus Bio-Medico, Rome
- Clatterbridge Centre for Oncology, Bebington, Wirral, United Kingdom